CLINICAL TRIAL: NCT00851448
Title: Safety, Tolerance and Efficacy of an Oral Nutritional Supplement in Lung Cancer Patients. A Randomised, Double-blind, Controlled Pilot Study
Brief Title: Safety, Tolerance and Efficacy of an Oral Nutritional Supplement in Lung Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Dr. Ericka Pestana, I&D Clinical Nutrition & Pharmaceuticals, SP&T, Fresenius Kabi Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PCSU-001-CFS
Record Dates: First submitted 2009-02-13; First posted 2009-02-26 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Cachexia; Cancer
MeSH Terms: conditions — Cachexia; Neoplasms | interventions — Dietary Supplements; Food

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Oral nutritional supplement containing n-3 fatty acids, amino acids, antioxidants
  Interventions: Dietary Supplement: oral nutritional supplement, food for special medical purposes
- 2 (Placebo Comparator): isocaloric, isonitrogenous
  Interventions: Dietary Supplement: oral nutritional supplement, food for special medical purposes

INTERVENTIONS:
Dietary Supplement: oral nutritional supplement, food for special medical purposes — 2 servings of 200-300 ml per day, treatment period: 16 weeks

SUMMARY:
To test the compliance, tolerance, safety and to get preliminary insights into the efficacy of a new oral nutritional supplement (containing n-3 fatty acids, amino acids and antioxidants) designed to prevent or delay cachexia and anorexia in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer patients stage IIIb or IV
* planned chemotherapy or combined chemo-/radiotherapy
* current body weight less than 6 months ago
* abnormal CRF level
* BMI >=20 kg/m2 and <=30kg/m2

Exclusion Criteria:

* significant oedema in the time of screening and randomisation
* concomitant inflammatory diseases
* active infections including HIV and AIDS
* liver failure
* chronic renal failure or cardiac pacemaker
* chronic heart failure
* insulin treated diabetes mellitus
* medications that impair sex hormone synthesis, secretion or function
* acute or chronic infections
* body weight loss > 5% during the last 6 months or > 10% during the last 10 months
* fish oil supplementation within 3 months prior to study entry
* taking vitamins in doses greater than recommended daily allowance
* life expectancy less than 6 months in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
compliance to nutrition therapy | baseline, months 1, 2, 3, 4

SECONDARY OUTCOMES:
anorexia questionnaire | baseline, months 1, 2, 3, 4
gastrointestinal syndrome score (GIS) | baseline, months 1, 2, 3, 4
body cell mass | baseline, months 1, 2, 3, 4
weight change | baseline, months 1, 2, 3, 4
hand grip strength | baseline, months 1, 2, 3, 4
ECOG performance status | baseline, months 1, 2, 3, 4

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Rossi-Fanelli, Professor, Principal Investigator — La Sapienza Università, Rome
Locations (3):
- Dipartimento di Medicina Clinica, La Sapienza Università, Rome, Rome, Italy
- Poland (2):
  - Indywidualna Specjalistyczna Praktyka lekarska, Ruda Śląska
  - Pulmonology Dept. of Miedzylesie Hospital, Warsaw